CLINICAL TRIAL: NCT07275294
Title: Combined Effects of Pelvic Floor Exercises and Muscle Energy Techniques on Pain and Functional Disability in Patients With Sacroiliac Joint Dysfunction: A Randomized Controlled Trial
Brief Title: Effects of Pelvic Floor Exercises and Muscle Energy Techniques on Pain and Disability in Sacroiliac Joint Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Tariq Rafiq, Associate Professor, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/027
Record Dates: First submitted 2025-11-21; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: Pain; Functional Disability; Pelvic floor exercises; Muscle energy techniques; Sacroiliac joint dysfunction
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Muscle Energy Techniques with Hot pack and Transcutaneous Electrical Nerve Stimulation
  Interventions: Other: Muscle Energy Techniques with Hot pack and Transcutaneous Electrical Nerve Stimulation
- Experimental Group (Experimental): Muscle Energy Techniques with Hot pack, Transcutaneous Electrical Nerve Stimulation and Pelvic Floor Exercises
  Interventions: Other: Muscle Energy Techniques with Hot pack, Transcutaneous Electrical Nerve Stimulation and Pelvic floor Exercises

INTERVENTIONS:
Other: Muscle Energy Techniques with Hot pack and Transcutaneous Electrical Nerve Stimulation — There will be an application of a hot pack for 10minutes and TENS for 10minutes. After that Muscle Energy Techniques (METs) will be performed as isometric relaxation technique targeting iliopsoas, piriformis, hamstring and gluteus medius muscles. The protocol will involve isometric contraction in which patients will perform a contraction at ~30% effort against the therapist's resistance for 7-10 seconds. A 5-second relaxation phase followed by a stretch to the new range barrier, held for 10-60 seconds. Each stretch will be repeated 3-5 in each session. This will be performed 3 times per session 3 times per week for 6 weeks.
  Arms: Control group
Other: Muscle Energy Techniques with Hot pack, Transcutaneous Electrical Nerve Stimulation and Pelvic floor Exercises — There will be an application of a hot pack for 10minutes and TENS for 10minutes. After that Muscle Energy Techniques (METs) will be performed as isometric relaxation technique targeting iliopsoas, piriformis, hamstring and gluteus medius muscles. The protocol will involve isometric contraction in which patients will perform a contraction at ~30% effort against the therapist's resistance for 7-10 seconds. A 5-second relaxation phase followed by a stretch to the new range barrier, held for 10-60 seconds. Each stretch will be repeated 3-5 in each session. This will be performed 3 times per session 3 times per week for 6 weeks.
  Participants in the experimental group will be instructed to perform the Pelvic Floor Exercises (Kegel exercises, Pelvic Tilts and Bridge with pelvic floor engagement) according to the defined protocol.
  Arms: Experimental Group

SUMMARY:
This clinical trial aims to evaluate whether combining pelvic floor exercises with muscle energy techniques provides greater improvement in pain and functional disability in adults with sacroiliac joint dysfunction compared to muscle energy techniques alone. The study examines whether the addition of pelvic floor training enhances pain reduction and functional outcomes beyond the effects of muscle energy techniques applied to the hamstrings, gluteus medius, piriformis, and iliopsoas muscles. Participants will be assigned to either an experimental group receiving both pelvic floor exercises and muscle energy techniques or a control group receiving muscle energy techniques only, and will complete standardized assessments of pain and disability before and after the intervention.

DETAILED DESCRIPTION:
This clinical trial is designed to evaluate the combined therapeutic effects of pelvic floor muscle exercises and muscle energy techniques on pain intensity and functional disability in individuals with sacroiliac joint dysfunction. It is commonly linked to altered lumbopelvic mechanics and impaired stability, and interventions that target both joint alignment and deep stabilizing musculature may offer improved clinical outcomes. All participants will undergo baseline assessment, including sacroiliac joint pain provocation tests, pain intensity measured with the Numeric pain rating scale, and functional disability assessed using the Modified Oswestry Disability Index. The intervention will occur three times per week for six weeks, with each session lasting approximately 40-45 minutes. Both groups will receive standard physiotherapy consisting of a hot pack and Transcutaneous Electrical Nerve Stimulation for pain modulation, followed by muscle energy techniques directed at the hamstrings, gluteus medius, piriformis, and iliopsoas to improve muscle balance and sacroiliac joint mobility. The experimental group will additionally participate in a structured pelvic floor exercise program designed to enhance pelvic stability and reinforce load transfer across the sacroiliac joint. Participants will be advised to avoid any external treatments during the study period. Post-intervention assessments will be conducted immediately, after three weeks of treatment and again at six weeks post-treatment to determine both immediate and short-term follow-up effects. This study aims to clarify whether the integration of pelvic floor exercises with traditional muscle energy techniques results in superior clinical outcomes compared to muscle energy techniques alone in the management of sacroiliac joint dysfunction.

ELIGIBILITY:
Inclusion Criteria

* Unilateral sacroiliac joint dysfunction pre diagnosed patients
* Both male and female
* Age 30 to 50 years
* Positive on at-least 3/5 provocation tests (Compression, Distraction, Gaenslen, Thigh Thrust, Sacral Thrust and FABER (Flexion, Abduction, External Rotation) test)
* Pain at Fortin area
* Symptoms >3 weeks

Exclusion Criteria:

* Pregnant females
* Any other neurological, orthopedic, or musculoskeletal disorder
* Recent history of pelvic surgery or any history of malignancy
* Lumbar pathologies (scoliosis, spondylosis, spondylolisthesis)
* Sacroiliitis

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain for SIJD provocation tests | From enrollment to the end of treatment at 6 weeks
  The NRS is a widely used, unidimensional tool for assessing pain intensity. It asks the individual to rate their pain on a scale of 0 (no pain) to 10 (worst pain imaginable). It is easy to understand and quick to administer and score. It is used for various types of pain (acute and chronic) and in different settings. The NPRS has demonstrated good to excellent reliability and validity with low back pain. Pain scores categorized as mild pain (1-3), moderate pain (1-3) and severe pain (7-10).

SECONDARY OUTCOMES:
Functional Disability | From enrollment to the end of treatment at 6 weeks
  Functional disability is measured using the Modified Oswestry Disability Index. It asks questions about everyday activities such as sitting, standing, walking, lifting, and personal care. The Modified Oswestry Disability Index is a patient-completed questionnaire that measures functional disability using 10 questions with 6-point Likert scales. Each question is scored from 0 (no disability) to 5 (maximum disability). The total Modified Oswestry Disability Index score is a percentage reflecting how much low back pain affects daily life. It is calculated by dividing the individual's score by the maximum possible score and converting it into a percentage. The resulting percentage falls into a category that indicates the level of disability. The participants experience mild pain and can perform most activities with a score of 0-20% (Minimal disability).The participants experience severe functional limitation with a score of 81-100% (bed-bound or exaggerating symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD TARIQ RAFIQ, PhD, Principal Investigator — Lahore University of Biological & Applied Sciences

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: It will be available after the completion of the study.
Access Criteria: Through the corresponding author.